CLINICAL TRIAL: NCT01051219
Title: A Randomised, Controlled Trial of Losartan as an Anti-fibrotic Agent in Non-alcoholic Steatohepatitis
Brief Title: Anti-Fibrotic Effects of Losartan In Nash Evaluation Study
Acronym: FELINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EME-08/43/15; ISRCTN (Registry Identifier: 57849521)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Losartan; Liver fibrosis; Nonalcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan, daily medication (Active Comparator): 50 milligrams Losartan to be taken orally daily
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): A matched placebo will be given for patients to take once daily
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — 50 milligrams to be taken orally, daily
  Other Names: Losartan also known as Cozaar

SUMMARY:
This is a randomized, controlled trial to determine whether Losartan is effective at slowing down, halting or reversing liver fibrosis in patients with non-alcoholic steatohepatitis (NASH). Liver fibrosis is the accumulation of tough, fibrous scar tissue in the liver which occurs in patients with NASH. NASH resembles alcoholic liver disease, but occurs in people who drink little or no alcohol. The major feature in NASH is fat in the liver, along with inflammation and damage, which may lead to cirrhosis, in which the liver is permanently damaged and scarred and no longer able to function properly.

Primary hypothesis:

That losartan is superior to placebo in reversing, slowing down or halting fibrosis in patients with non-alcoholic fatty liver disease, after 24 months of treatment.

Secondary hypothesis:

1. That the safety profile of the angiotensin receptor blocker (losartan) in this patient population is acceptable
2. That losartan can prevent clinical deterioration in non-alcoholic fatty liver disease
3. That serum, radiological and histological markers of fibrosis correlate in these patients over a 24 month period

ELIGIBILITY:
Inclusion Criteria:

* Adults (both males and females, aged 18+) with steatohepatitis and fibrosis (Kleiner F1-F3), resulting from non-alcoholic fatty liver disease.

Exclusion Criteria:

* Refusal or inability (lack of capacity) to give informed consent
* Average alcohol ingestion >21 units/week (males) or >14 units/week (females)
* History or presence of Type 1 diabetes mellitus
* Haemoglobin A1C >15.0
* Other causes of chronic liver disease or hepatic steatosis
* Any contra-indication to liver biopsy
* History of, or planned, gastrointestinal bypass surgery
* Hepatocellular carcinoma
* Previous liver transplantation
* Recent significant weight loss (>5% total body weight within last 6 months)
* Electrolyte disturbance: potassium level outside the normal (local) range
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >10 x upper limit of normal (ULN) at screening
* Recent (within 6 months of baseline liver biopsy and screening visit) or concomitant use of agent known to cause hepatic steatosis (corticosteroids, amiodarone, methotrexate, tamoxifen, tetracycline, high dose oestrogens, valproic acid), or concomitant use of pioglitazone, fluconazole, rifampicin or any drug contra-indicated in the Losartan SmPC
* Introduction of metformin, glitazones, a GLP-1 agonist, Vitamin E or C, betaine, s-adenosyl methionine, ursodeoxycholic acid, silymarin, fibrate, pentoxifylline, orlistat, sibutramine or rimonabant within 3 months of baseline liver biopsy and screening visit
* Intolerance of angiotensin receptor blockers (ARBs) or presence of multiple allergic reactions to drugs
* Use of angiotensin-converting enzyme (ACE) inhibitor or ARB in previous year
* Hypotension (systolic <100, diastolic <60)
* Renal failure (Cr >130)
* Participation in any clinical study of an investigational agent within 30 days or five half-lives of the investigational product, whichever is longer
* Presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, haematological, neurological, psychiatric, systemic, ocular, gynaecologic or any acute infectious disease or signs of acute illness that, in the opinion of the investigator, might compromise the patient's safe participation in the trial
* Presence or history of cancer within the past 5 years with exception of adequately treated localized basal cell carcinoma of the skin, in situ cervical carcinoma or solid malignancy surgically excised in toto without recurrence for five years
* Women of child-bearing potential not protected by effective contraceptive method of birth control or surgical sterilization and/or who are unwilling or unable to be tested for pregnancy (Pregnancy status will be checked by serum pregnancy testing before initiation of study treatment and by urine pregnancy testing during the trial)
* Known allergy or sensitivity to losartan or its excipients (microcrystalline cellulose [E460]; lactose monohydrate; pregelitanized maize starch; magnesium stearate [E572]; hydroxypropyl cellulose [E463]; hypromellose [E464])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be change in Kleiner fibrosis score, [Kleiner DE et al Hepatology 2005], based on histological fibrosis stage (as judged by two independent blinded histopathologists from liver biopsies), from pre-treatment to end-of-study | trial entry, end of study (2 years)

SECONDARY OUTCOMES:
Change in radiological (fibroscan) and serological (ELF) markers of fibrosis | trial entry, 48 weeks, 96 weeks
change in NAFLD activity score (NAS) | trial entry, end of study
comparison of "responder rate" - placebo versus intervention | trial entry, end of study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Day, PhD, Study Chair — Newcastle University; Derek Mann, PhD, Study Director — Newcastle University; Stephen F Stewart, PhD, Study Director — Newcastle University; Elaine McColl, PhD, Study Director — Newcastle University; Ian N Steen, PhD, Study Director — Newcastle University
Locations (10):
- United Kingdom (10):
  - Plymouth Hospitals NHS Trust, Plymouth, Devon
  - Queen Elizabeth Hospital, Birmingham
  - Cambridge University NHS Foundation Trust, Cambridge
  - Royal Derby Hospital, Derby
  - Royal Liverpool & Broadgreen University Hospital, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College (St Mary's Site), London
  - St George's Hospital, London
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Queens Medical Centre, Nottingham

REFERENCES:
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Newton JL, Jones DE, Henderson E, Kane L, Wilton K, Burt AD, Day CP. Fatigue in non-alcoholic fatty liver disease (NAFLD) is significant and associates with inactivity and excessive daytime sleepiness but not with liver disease severity or insulin resistance. Gut. 2008 Jun;57(6):807-13. doi: 10.1136/gut.2007.139303. Epub 2008 Feb 12. PMID 18270241
- [Background] Lindor KD, Kowdley KV, Heathcote EJ, Harrison ME, Jorgensen R, Angulo P, Lymp JF, Burgart L, Colin P. Ursodeoxycholic acid for treatment of nonalcoholic steatohepatitis: results of a randomized trial. Hepatology. 2004 Mar;39(3):770-8. doi: 10.1002/hep.20092. PMID 14999696
- [Background] Adams LA, Sanderson S, Lindor KD, Angulo P. The histological course of nonalcoholic fatty liver disease: a longitudinal study of 103 patients with sequential liver biopsies. J Hepatol. 2005 Jan;42(1):132-8. doi: 10.1016/j.jhep.2004.09.012. PMID 15629518
- [Background] Adams LA, Lymp JF, St Sauver J, Sanderson SO, Lindor KD, Feldstein A, Angulo P. The natural history of nonalcoholic fatty liver disease: a population-based cohort study. Gastroenterology. 2005 Jul;129(1):113-21. doi: 10.1053/j.gastro.2005.04.014. PMID 16012941
- [Background] Wright MC, Issa R, Smart DE, Trim N, Murray GI, Primrose JN, Arthur MJ, Iredale JP, Mann DA. Gliotoxin stimulates the apoptosis of human and rat hepatic stellate cells and enhances the resolution of liver fibrosis in rats. Gastroenterology. 2001 Sep;121(3):685-98. doi: 10.1053/gast.2001.27188. PMID 11522753
- [Background] Watson MR, Wallace K, Gieling RG, Manas DM, Jaffray E, Hay RT, Mann DA, Oakley F. NF-kappaB is a critical regulator of the survival of rodent and human hepatic myofibroblasts. J Hepatol. 2008 Apr;48(4):589-97. doi: 10.1016/j.jhep.2007.12.019. Epub 2008 Jan 31. PMID 18279996
- [Background] Oakley F, Meso M, Iredale JP, Green K, Marek CJ, Zhou X, May MJ, Millward-Sadler H, Wright MC, Mann DA. Inhibition of inhibitor of kappaB kinases stimulates hepatic stellate cell apoptosis and accelerated recovery from rat liver fibrosis. Gastroenterology. 2005 Jan;128(1):108-20. doi: 10.1053/j.gastro.2004.10.003. PMID 15633128
- [Background] Bataller R, Sancho-Bru P, Gines P, Lora JM, Al-Garawi A, Sole M, Colmenero J, Nicolas JM, Jimenez W, Weich N, Gutierrez-Ramos JC, Arroyo V, Rodes J. Activated human hepatic stellate cells express the renin-angiotensin system and synthesize angiotensin II. Gastroenterology. 2003 Jul;125(1):117-25. doi: 10.1016/s0016-5085(03)00695-4. PMID 12851877
- [Background] Bataller R, Gabele E, Parsons CJ, Morris T, Yang L, Schoonhoven R, Brenner DA, Rippe RA. Systemic infusion of angiotensin II exacerbates liver fibrosis in bile duct-ligated rats. Hepatology. 2005 May;41(5):1046-55. doi: 10.1002/hep.20665. PMID 15841463